CLINICAL TRIAL: NCT06713018
Title: Prospective, Multicenter, Randomized Controlled Clinical Study of Orthopedic Intelligent Navigation System in the Treatment of Fresh Femoral Neck Fractures
Brief Title: Orthopedic Intelligent Navigation System in the Treatment of Fresh Femoral Neck Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhang Wei, Deputy head of orthopedics, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2024-341-01
Record Dates: First submitted 2024-11-16; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Fracture of Neck of Femur
Keywords: orthopedic intelligent navigation system
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three cannulated compression screws by navigation system (Experimental)
  Interventions: Procedure: Three cannulated compression screws by navigation system
- Traditional three cannulated compression screws (Placebo Comparator)
  Interventions: Procedure: Traditional three cannulated compression screws

INTERVENTIONS:
Procedure: Three cannulated compression screws by navigation system — Patients with femoral neck fractures treated with three cannulated compression screws assisted by a navigation system
  Arms: Three cannulated compression screws by navigation system
Procedure: Traditional three cannulated compression screws — Patients with femoral neck fractures treated with traditional three cannulated compression screws
  Arms: Traditional three cannulated compression screws

SUMMARY:
The goal of this clinical trial is to verify the safety and effectiveness of orthopaedic surgical navigation system in the treatment of fresh femoral neck fractures.

Participants will:

* Take three cannulated compression screws by navigation system or by traditional method to treat femoral neck fractures.
* Visit the clinic 1, 3, 6, 12 months after surgery for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender is not limited;
2. Patients diagnosed with femoral neck fracture;
3. Patients with indications for internal fixation of femoral neck fracture and able to tolerate surgery;
4. The subject or his legal representative is informed of the nature of the study and agrees to participate in the study.

Exclusion Criteria:

1. Participants who had participated in clinical studies of other drugs, biologics or medical devices before enrollment and did not reach the primary study endpoint time limit;
2. The patient is known to have a history of allergy to one or more implanted materials;
3. Patients determined by researchers to be physically weak or unable to tolerate surgery due to other systemic diseases;
4. Active infection of the hip joint or other parts of the body is determined by the investigator;
5. Diagnosed as metabolic bone disease, radiation bone disease, etc.;
6. Severe hip contracture deformity or severe muscle loss fused to the functional position for a long time without pain;
7. have inflammatory arthritis, such as rheumatoid arthritis, systemic lupus erythematosus arthritis, ankylosing spondylitis, etc.;
8. The patient is mentally incapable or unable to understand the requirements of participating in the study, and it is difficult to cooperate;
9. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Perspective frequency | 1 day
  Document the total number of intraoperative fluoroscopy sessions taken during surgery, including each anteroposterior and lateral fluoroscopic image

SECONDARY OUTCOMES:
Neck shaft angle | 1 year
Guide needle implantation effect | 1 day
  For the group treated with three hollow compression screws, the effect of the implantation of guide pins is categorized into three parallel pins, two parallel pins, and mutually non-parallel pins, with measurements taken during the surgery.
Fluoroscopy times of needle implantation | 1 day
Operation time | 1 day
Operative blood loss | 1 day
Fracture union | 1 year
  Postoperative follow-up observation is conducted for all patients, with anteroposterior and lateral hip X-rays taken at the 1st, 3rd, 6th, and 12th postoperative months. X ray and CT scans are reviewed at the 1st and 3rd postoperative months to observe the stability of the implanted internal fixation, the disappearance of the fracture line, and whether there is displacement of the fracture ends.
Zarit Burden Interview score | 1 year
  The Zarit Burden Interview (ZBI) is a commonly used assessment tool designed to quantify the psychological and emotional burden experienced by caregivers who provide care for individuals with cognitive or functional impairments. Developed by Zarit and colleagues, the scale consists of 22 items that cover various aspects of caregiver burden, such as time pressure, emotional strain, and social isolation. The scoring ranges from 0 to 88, with higher scores indicating a greater level of caregiving burden. This tool aids healthcare professionals in identifying the psychological stress faced by caregivers and provides appropriate support and interventions to improve their mental health and quality of life.
Harris score | 1 year
  The Harris Score (Harris Hip Score, HHS) is a widely used scale for evaluating hip joint function and patient quality of life, often applied to assess the outcomes of hip replacement surgery or other treatments for hip joint diseases. It covers four main aspects: pain level, functional activity, joint range of motion, and hip joint deformity. The total score ranges from 0 to 100, with 100 being the best possible condition, indicating complete normalcy of hip joint function.
SF-36 score | 1 year
  The SF-36 (Short Form 36 Health Survey) is a widely used generic health status assessment tool developed by the Medical Outcomes Study (MOS) Group. The scale is designed to comprehensively evaluate health-related quality of life, encompassing eight dimensions: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, bodily pain, mental health, vitality, and general health perceptions. Each dimension consists of several items, and scores are derived by summing the scores of these items, typically converted to a 0 to 100 percent scale, with 100 representing the best possible health state. These eight dimension scores can be combined to form two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No